CLINICAL TRIAL: NCT00064090
Title: A Phase I Study of Triapine and Cytarabine in Patients With Hematologic Malignancies
Brief Title: 3-AP and Cytarabine in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: VION-CLI-032; CDR0000306465 (Registry Identifier: PDQ (Physician Data Query)); MDA-DM-030096
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2008-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; blastic phase chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; relapsing chronic myelogenous leukemia; chronic myelomonocytic leukemia; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; previously treated myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Blast Crisis; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — Cytarabine; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

INTERVENTIONS:
Drug: cytarabine
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as cytarabine use different ways to stop cancer cells from dividing so they stop growing or die. 3-AP may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth and may help cytarabine kill more cancer cells by making them more sensitive to the drug.

PURPOSE: Phase I trial to study the effectiveness of combining cytarabine with 3-AP in treating patients who have relapsed or refractory hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility, tolerability, and toxic effects of 3-AP in combination with cytarabine in patients with hematologic malignancies.
* Determine the maximum tolerated dose and phase II dose of cytarabine in this regimen in these patients.
* Determine the biological effects of 3-AP and its interaction with cytarabine in these patients.

OUTLINE: This is a pilot, dose-escalation study of cytarabine.

Patients receive 3-AP IV over 6 hours followed by cytarabine IV over 18 hours on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a response may receive an additional course as consolidation therapy.

Cohorts of 3-6 patients receive escalating doses of cytarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 10 patients receive treatment at that dose.

PROJECTED ACCRUAL: Approximately 20-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Acute myeloid leukemia
  * Acute lymphoblastic leukemia
  * Chronic myelogenous leukemia (CML)
  * CML in blast crisis
  * Chronic lymphocytic leukemia
  * High-risk* myelodysplastic syndromes, including the following:

    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
    * Chronic myelomonocytic leukemia NOTE: *High-risk myelodysplasia defined as having an International Performance Scoring System score of at least 1.5, based on adverse cytogenetics, greater than 10% blasts in marrow, and cytopenias in at least 2 lineages
* Relapsed or refractory disease
* Ineligible for higher priority protocols

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 2 months

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin no greater than 2.0 mg/dL (unless considered due to malignancy)
* ALT or AST no greater than 3 times upper limit of normal
* Chronic hepatitis allowed

Renal

* Creatinine no greater than 2.0 mg/dL (unless considered due to malignancy)

Cardiovascular

* No myocardial infarction within the past 3 months
* No symptomatic coronary artery disease
* No arrhythmias (other than atrial fibrillation or flutter) requiring treatment
* No uncontrolled congestive heart failure

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Concurrent infections under active treatment with and controlled by antibiotics allowed
* No other concurrent life-threatening illness
* No mental deficit or psychiatric history that would preclude giving informed consent or complying with protocol

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 1 week since prior growth factors, including the following:

  * Epoetin alfa
  * Filgrastim (G-CSF)
  * Sargramostim (GM-CSF)
  * Interleukin-3
  * Interleukin-11
* No concurrent anticancer immunotherapy

Chemotherapy

* At least 72 hours since prior hydroxyurea
* Recovered from prior chemotherapy
* No other concurrent anticancer chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 2 weeks since prior radiotherapy
* No concurrent anticancer radiotherapy

Surgery

* Not specified

Other

* At least 3 weeks since prior myelosuppressive cytotoxic agents (in the absence of rapidly progressing disease)
* At least 1 week since prior nonmyelosuppressive therapy
* No other concurrent standard or investigational therapy for the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03; Primary Completion 2004-09 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States